CLINICAL TRIAL: NCT04172155
Title: Effects of Pulmonary Rehabilitation on Self-esteem in Patients With COPD
Brief Title: Pulmonary Rehabilitation and Self-esteem in Patients With COPD
Acronym: ESMOI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ESMOI (29BRC19.0225)
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the aim of this study is to evaluate the evolution of self-esteem during a pulmonary rehabilitation program, in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage 2 to 4 (A to D) COPD admitted to a pulmonary rehabilitation program
* Patient aged 18 or over
* Patient able to consent and having signed a consent form

Exclusion Criteria:

* Patient with pain, osteoarthritis or shoulder surgery
* Patient with a history of Pneumonectomy, lobectomy less than 6 months old
* Refusal of participation
* Patient with an inability to complete a pulmonary rehabilitation program in totality
* Pregnant or breast-feeding women
* Patient under tutorship or curatorship

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted to a pulmonary rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
PSI-6 | PSI-6 is measured at the biginning and at the end of the pulmonary rehabilitation program (4 weeks)
  the physical self inventory- 6 (PSI-6) allows to evaluate self esteem

SECONDARY OUTCOMES:
6MWT | the 6MWT is measured at the biginning and at the end of the pulmonary rehabilitation program (4 weeks)
  The 6-minute walk test allows to evaluate exercise capacity
HAD | HAD is measured at the biginning and at the end of the pulmonary rehabilitation program (4 weeks)
  the hospital anxiety and depressive scale (HAD) measure the anxiety and depression
SGRQ | SGRQ is measured at the biginning and at the end of the pulmonary rehabilitation program (4 weeks)
  the Saint-George respiratory Questionnaire (SGRQ) measure the quality of life

OTHER OUTCOMES:
MMRC | MMRC is measured at the biginning and at the end of the pulmonary rehabilitation program (4 weeks)
  The modified medical research Council dyspnea scale measure dyspnea

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CH Pays de Morlaix, Morlaix

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Fox, K.R. et Corbin, C.B.The Physical Self-Perception Profile : Devlopment and Preliminary Validation. Journal of Sport and Exercise Psychology, 11(4), p. 408 430, 1989
- [Background] Ninot G, Moullec G, Desplan J, Prefaut C, Varray A. Daily functioning of dyspnea, self-esteem and physical self in patients with moderate COPD before, during and after a first inpatient rehabilitation program. Disabil Rehabil. 2007 Nov 30;29(22):1671-8. doi: 10.1080/09638280601055949. PMID 17852227